CLINICAL TRIAL: NCT00944970
Title: Vasodilator Induced Stress In CONcordance With Adenosine (VISION-305)
Brief Title: Efficacy and Safety Study of Binodenoson in Assessing Cardiac Ischemia
Acronym: VISION-305
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MRE0470P-305
Record Dates: First submitted 2009-07-17; First posted 2009-07-23 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Angina; Anginal symptoms; Ischemic heart disease; Ischemia; Single photon emission computed tomography; Pharmacologic stress; Myocardial perfusion imaging; Suspected coronary artery disease; known coronary artery disease; typical or atypical anginal symptoms
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Ischemia; Ischemia | interventions — binodenoson; Adenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- binodenoson then adenosine (Other): binodenoson (experimental); adenosine (active comparator)
  Interventions: Drug: binodenoson; Drug: adenosine
- adenosine then binodenoson (Other): adenosine (active comparator); binodenoson (experimental)
  Interventions: Drug: binodenoson; Drug: adenosine
- adenosine then adenosine (Active Comparator)
  Interventions: Drug: adenosine

INTERVENTIONS:
Drug: binodenoson — 30-second intravenous injection (bolus) of binodenoson (1.5 mcg/kg) and a 6-minute intravenous infusion of placebo
  Other Names: CorVue
  Arms: adenosine then binodenoson; binodenoson then adenosine
Drug: adenosine — 30-second intravenous injection (bolus) of placebo and a 6-minute intravenous infusion of adenosine (140 mcg/kg/minute)

SUMMARY:
Binodenoson (an experimental drug) and adenosine (an FDA-approved drug that is currently used by doctors) are used to increase blood flow to the heart just like when a person exercises on a treadmill. Using imaging techniques, this increased blood flow can help determine if areas of the heart are not getting enough blood and oxygen during exercise. The purpose of the study is to determine if binodenoson is as good as adenosine in determining if there are areas of the heart not getting enough oxygen when blood flow to the heart is increased.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an informed consent form.

Exclusion Criteria:

* Women who are of childbearing potential.
* Very low likelihood of coronary artery disease (by American Heart Association and American College of Cardiology standards).
* Documented history of acute myocardial infarction within 30 days.
* Percutaneous coronary intervention or coronary bypass graft surgery within 3 years, unless typical or atypical anginal symptoms are present.
* Reactive airway disease or other contraindication that preclude a patient from receiving adenosine.
* Previous heart transplant or listed to receive a heart transplant.
* Cardiomyopathy (idiopathic dilated, restrictive, hypertrophic).
* History of hemodynamically significant supraventricular tachycardia or sustained ventricular tachycardia.
* Presence of second- or third-degree AV block (in the absence of permanent pacemaker).
* Left ventricular ejection fraction greater than 35%, known prior to the first imaging procedure.
* Presence of advanced heart failure, New York Heart Association Class IV.
* History of vasospastic/Prinzmetal angina.
* Active (under treatment) cancer (except skin cancers).
* Inability to discontinue antianginal medications, Aggrenox®, dipyridamole, and xanthine-containing drugs and foods (including caffeine) as required prior to each imaging procedure.
* Previous participation in a study of binodenoson.
* Any physical or psychosocial condition that, based on the Investigator's judgment, would prevent the patient from completing the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2005-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Summed difference in binodenoson and adenosine reader-generated Summed Difference Scores | 2 to 7 days apart
Summed difference in adenosine- and adenosine-2 reader-generated Summed Difference Scores | 2 to 7 days apart
Extreme discrepancies in binodenoson and adenosine reader-generated Summed Difference Scores | 2 to 7 days apart
Extreme discrepancies in adenosine- and adenosine-2 reader-generated Summed Difference Scores | 2 to 7 days apart

SECONDARY OUTCOMES:
Categorized reader-generated Summed Difference Scores (binodenoson and adenosine) | 2 to 7 days apart
Categorized reader-generated Summed Difference Scores (adenosine-1 and adenosine-2) | 2 to 7 days apart
Difference in reader-generated Summed Stress Scores (binodenoson and adenosine) | 2 to 7 days apart
Difference in reader-generated Summed Stress Scores (adenosine-1 and adenosine-2) | 2 to 7 days apart
Extreme discrepant reader-generated Summed Stress Scores (binodenoson and adenosine) | 2 to 7 days apart
Extreme discrepant reader-generated Summed Stress Scores (adenosine-1 and adenosine-2) | 2 to 7 days apart
Categorized reader-generated Summed Stress Scores (binodenoson and adenosine) | 2 to 7 days apart
Categorized reader-generated Summed Stress Scores (adenosine-1 and adenosine-2) | 2 to 7 days apart
Sensitivity compared to coronary angiography | angiography obtained up to 60 days post-image
Specificity compared to coronary angiography | angiography obtained up to 60 days post-image
Sensitivity compared to clinical endpoint | clinical endpoint obtained up to 60 days post-image
Specificity compared to clinical endpoint | clinical endpoint obtained up to 60 days post-image
Incidence of second- or third-degree AV block | 0 to 60 minutes after start of study drug administration
Patient-rated overall symptom bother | 1 hour post-dosing
Patient preference for pharmacologic stress agent | 1 to 4 days following 2nd procedure
Incidence of flushing | 0 to 60 minutes after start of study drug administration
Patient-rated intensity of flushing | 0 to 60 minutes after start of study drug administration
Incidence of chest pain | 0 to 60 minutes after start of study drug administration
Patient-rated intensity of chest pain | 0 to 60 minutes after start of study drug administration
Incidence of dyspnea | 0 to 60 minutes after start of study drug administration
Patient-rated intensity of dyspnea | 0 to 60 minutes after start of study drug administration
Incidence of nausea | 0 to 60 minutes after start of study drug administration
Patient-rated intensity of nausea | 0 to 60 minutes after start of study drug administration
Incidence of headache | 0 to 60 minutes after start of study drug administration
Patient-rated intensity of headache | 0 to 60 minutes after start of study drug administration
Incidence of abdominal discomfort | 0 to 60 minutes after start of study drug administration
Patient-rated intensity of abdominal discomfort | 0 to 60 minutes after start of study drug administration
Incidence of dizziness | 0 to 60 minutes after start of study drug administration
Patient-rated intensity of dizziness | 0 to 60 minutes after start of study drug administration
Overall incidence of adverse events | up to 7 days post-dosing
Peak change in heart rate | 0 to 60 minutes after start of study drug administration
Peak change in systolic blood pressure | 0 to 60 minutes after start of study drug administration
Peak change in diastolic blood pressure | 0 to 60 minutes after start of study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Rolleri, Pharm.D., Study Director — King Pharmaceuticals is now a wholly owned subsidiary of Pfizer